STUDY: Perioperative Ketamine in Opioid-Tolerant Patients Undergoing Lumbar Spine Surgery: A

Randomized, Double-blind, Place-controlled Trial

Principal Investigator: Jacques E. Chelly, MD, PhD, MBA

**IRB:** STUDY19020144

**NCT:** 04220489

Statistical Analysis Plan – Approved 09/03/2019

This is a pilot to support a P01 program pilot application to the NIH, so the data will be analyzed mainly using descriptive statistics. Additional statistical analysis methods such as a 2-sample t test to compare significance between groups may also occur.